CLINICAL TRIAL: NCT04430790
Title: Doxapram Versus Placebo in Preterm Newborns: An International Double Blinded Multicenter Randomized Controlled Trial
Brief Title: Doxapram Therapy in Preterm Infants (DOXA Trial)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Nederlands Neonataal Netwerk (N3), the Netherlands (Unknown); Universitaire Ziekenhuizen KU Leuven (Other); Maternal, Infant, Child and Youth Research Network (MICYRN) (Unknown)
Responsible Party: Principal Investigator, Sinno H.P. Simons, Principal investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL72125.078.19; 80-84800-9843009 (Other Grant/Funding Number: ZonMw GGG); 2019-003666-41 (EudraCT Number)
Record Dates: First submitted 2020-01-08; First posted 2020-06-12 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Apnea of Prematurity; Respiratory Insufficiency
Keywords: Preterm infants; Hypoxia; Doxapram
MeSH Terms: conditions — Apnea; Respiratory Insufficiency; Hypoxia | interventions — Doxapram

STUDY DESIGN:
Intervention Model Description: Doxapram versus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxapram (Experimental): Blinded doxapram (2mg/ml, in glucose 5%) loading dose of 2.0 to 2.5 mg/kg administered in 5 to 10 minutes, followed by a continuous infusion of 0.5 - 1.0 mg/kg/hr ('www.kinderformularium.nl') as long as needed. Therapy is down titrated or stopped based on the patients' respiratory condition. If endotracheal intubation is needed study drug is stopped. After extubation study drug may be restarted. Switch to gastro-enteral administration is allowed if no iv-access is needed for other reasons.
  Interventions: Drug: Doxapram
- Placebo (Placebo Comparator): Placebo (glucose 5%) will also be administered with a loading dose and continuous infusion (in equal amounts of fluid as in experimental arm) by intravenous or gastro-intestinal infusion. The treatment protocol will be equal to the protocol in the doxapram arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxapram — Loading dose and continuous doxapram infusion.
  Other Names: Dopram
  Arms: Doxapram
Drug: Placebo — Loading dose and continuous placebo infusion.
  Other Names: Placebo (for Doxapram)
  Arms: Placebo

SUMMARY:
Preterm infants often suffer from apnea of prematurity (AOP; a cessation of breathing) due to immaturity of the respiratory system. AOP can lead to oxygen shortage and a low heart rate which might harm the development of the newborn, especially the central nervous system. In order to prevent oxygen shortage, infants are treated with non-invasive respiratory support and caffeine. Despite these treatments, many preterm newborns still suffer from AOP and need invasive mechanical ventilation. Although this will result in complete resolution of AOP, invasive mechanical ventilation has the disadvantage of being a major risk of chronic lung disease and impaired neurodevelopmental outcome. Restrictive invasive ventilation is therefore advocated nowadays in preterm infants. Doxapram is a respiratory stimulant that has been administered off-label to treat AOP. Doxapram, as add-on treatment, seems to be effective in treating AOP and to prevent invasive mechanical ventilation. It is unclear if a preterm infant benefit from doxapram treatment on the longer term. This study compares doxapram to placebo and hypothesizes that doxapram will protect preterm infants from both invasive ventilation (and related lung disease) and AOP related oxygen shortage (and related impaired brain development).

DETAILED DESCRIPTION:
The main objective of the trial is to investigate if doxapram is safe and effective in reducing the composite outcome of death and neurodevelopmental impairment/severe disability at 2 years corrected age as compared to placebo. This multicenter double blinded randomized placebo-controlled superiority trial will be conducted in multiple neonatal intensive care units in the Netherlands and Belgium, including 8 years follow-up. After written informed-consent the patients will be randomized into the doxapram treatment group or the placebo treatment group. Randomization will be stratified based on center and gestational age < or >= 26 weeks.

The participating departments include Dutch and Belgian Neonatal Intensive care units. The units include both academic and non-academic level III and IV units that are specialized in the care for critically ill and preterm born infants. Postnatal ages of patients at doxapram start vary from directly after birth up to months for the most-preterm born infants.

Blinded continuous doxapram or placebo (glucose 5%) will be infused as long as needed. Therapy is down titrated or stopped based on the patients' condition. If endotracheal intubation is needed study drug is stopped. After extubation study drug may be restarted. Switch to gastro-enteral administration is allowed if no iv-access is needed for other reasons. Next to study drug infusion, there will be no other study-related interventions. All outcome variables are already collected as standard of care. In a subset of patients doxapram plasma levels will be determined to validate the doxapram pharmacokinetic (PK) model. Blood will only be collected during routine blood sampling, with a maximum amount of 0.6 ml. Economic and cost-effectiveness evaluation will be performed. The national protocol for preterm birth advices follow-up at 2, 5.5 and 8 years respectively, as in the current study. Additional questionnaires will be used to collect data on the quality of life of patients and their parents.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the neonatal intensvie care unit (NICU) of one of the participating centres
* Written informed consent of both parents or legal representatives
* Gestational age at birth < 29 weeks
* Caffeine therapy, adequately dosed (see also under co-medication)
* Optimal Non-invasively supported with nasal Continuous Positive Airway Pressure (CPAP) or ventilation ((S)NIPPV, NIV-NAVA, BIPAP/Duopap, SIPAP)
* Apnea that require a medical intervention as judged by the attending physician

Exclusion Criteria:

* Previous use of open label doxapram
* Use of theophylline (to replace doxapram)
* Chromosomal defects (e.g. trisomy 13, 18, or 21)
* Major congenital malformations that: compromise lung function (e.g. surfactant protein deficiencies, congenital diaphragmatic hernia); result in chronic ventilation (e.g. Pierre Robin sequence); increase the risk of death or adverse neurodevelopmental outcome (congenital cerebral malformations, chromosomal abnormalities);
* Palliative care or treatment limitations because of high risk of impaired outcome.

Ages: 23 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 396 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2034-05-01 (Estimated)

PRIMARY OUTCOMES:
Death or severe disability | 2 years corrected age
  Disability will be defined as cognitive delay, cerebral palsy, severe hearing loss, or bilateral blindness. Cognitive delay will be defined as a Mental Development Index score of less than 85 on the Bayley Scales of Infant and Toddler Development, Bayley Score of Infant Development (BSID) III scores. Cerebral palsy will be diagnosed if the child had a non-progressive motor impairment characterized by abnormal muscle tone and decreased range or control of movements. The level of gross motor function will be determined with the use of the Gross Motor Function Classification System. Audiometry will be performed to determine the presence or absence of hearing loss. Blindness will be defined as a corrected visual acuity less than 20/200

SECONDARY OUTCOMES:
Broncho pulmonary dysplasia | 36 weeks post menstrual age
  Diagnosed according to the National Institute of Child Health and Human Development (NICHD) criteria
Death | until 36 weeks post menstrual age and until hospital discharge
  Death at 36 weeks post menstrual age and hospital mortality
Admission period | through study completion and until discharge home, average 3 months
  Length of stay at the intensive care, length of stay in hospital
Endotracheal intubations | Day 3, 7, 14, and 21 after start of study medication
  Incidence of endotracheal intubations
Oxygenation days and complications | During first hospital admittance and through study completion, average of 3 months
  Number of days on invasive ventilation, number of days on ventilatory support (non-invasive ventilation, CPAP, humidified high flow, low flow), number of days with supplemental oxygen, respiratory complications (airleak, pneumonia, etc), use of (rescue) corticosteroids for respiratory reasons.
Gastro-intestinal outcome measures | During first hospital admittance and until 36 weeks post menstrual age
  solitary intestinal perforation, necrotizing enterocolitis > stage 2 according to Bell, feeding problems with need for parental feeding (days with parental feeding after inclusion), body weight (gain, length), head circumference
Neurological outcome measures | During first hospital admittance or at term equivalent age (37-42 weeks postmenstrual age), average 3 months
  Intraventricular hemorhage(IVH) (all grades, grade III-IV, venous infarction), clinical seizures, periventricular leucomalacia (PVL) > gr 1)
Complications during neonatal period | During first hospital admittance or at term equivalent age (37-42 weeks postmenstrual age), average 3 months
  Incidence of late onset sepsis (culture proven or clinical suspected) and meningitis after inclusion, need for inotropes/circulatory support
Retinopathy of prematurity | During first hospital admittance or at term equivalent age (37-42 weeks postmenstrual age), average 3 months
  Grade of retinopathy (including plus disease and need for therapy)
Hearing | At term equivalent age, 37-42 weeks postmenstrual age, average 3 months
  Hearing test
Additional long term outcomes | 2 years corrected age
  Readmissions since first discharge home, weight/length/head circumference, behavioral problems (Child Behavior Checklist)
Parent reported outcome | 2 years corrected age
  Parent reported outcome with the PARCA-R (Parent Report of Children's Abilities-Revised) questionnaire (expected mean standardised scores 100 (SD 15), higher score is better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Smits, MD, PhD, Principal Investigator — Universitair Ziekenhuis Leuven; Karel Allegaert, MD, PhD, Study Director — Universitair Ziekenhuis Leuven
Locations (24):
- Belgium (10):
  - St Luc Louvain, Brussels, Avenaue Hippocrate 10
  - Delta Hospital Brussels, Brussels, Brussels Capital
  - University Hospital Brussels, Jette, Brussels Capital
  - Grand Hospital de Charleroi, Charleroi, Henegouwen
  - Clinique Saint-Vincent Liege, Liège, Liege
  - Academisch Ziekenhuis Sint-Jan, Bruges, West-Vlaanderen
  - Sint Augustinus Hospital Antwerp, Antwerp
  - University Hospital Antwerp, Antwerp
  - Chirec-Delta Hospital, Brussels
  - University Hospitals Leuven, Leuven
- Canada (5):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - McMaster Children's Hospital, Hamilton, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - Centre Mère-Enfent Soleil, Québec, Quebec
- Netherlands (9):
  - Radboudumc Amalia Children's Hospital Nijmegen, Nijmegen, Gelderland
  - Maastricht University Medical Center, Maastricht, Limburg
  - Maxima Medical Center Veldhoven, Veldhoven, North Brabant
  - Amsterdam University Medical Center, Amsterdam, North Holland
  - Isala Clinics Zwolle, Zwolle, Overijssel
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus Medical Center - Sophia Children's Hospital, Rotterdam, South Holland
  - University Medical Center Groningen, Groningen
  - UMC Utrecht - Wilhelmina Kinderziekenhuis, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: study protocol, sap and icf will be available at start of recruitment
Access Criteria: data will be available on request. Requests will be discussed by the steering committee
URL: https://dmp.radboudumc.nl/plans/31885/export.pdf?export%5Bquestion_headings%5D=true

REFERENCES:
- [Background] Poppe JA, Flint RB, Smits A, Willemsen SP, Storm KK, Nuytemans DH, Onland W, Poley MJ, de Boode WP, Carkeek K, Cassart V, Cornette L, Dijk PH, Hemels MAC, Hermans I, Hutten MC, Kelen D, de Kort EHM, Kroon AA, Lefevere J, Plaskie K, Stewart B, Voeten M, van Weissenbruch MM, Williams O, Zonnenberg IA, Lacaze-Masmonteil T, Pas ABT, Reiss IKM, van Kaam AH, Allegaert K, Hutten GJ, Simons SHP. Doxapram versus placebo in preterm newborns: a study protocol for an international double blinded multicentre randomized controlled trial (DOXA-trial). Trials. 2023 Oct 10;24(1):656. doi: 10.1186/s13063-023-07683-5. PMID 37817255